CLINICAL TRIAL: NCT01185275
Title: A Prospective Observational Study of Biopredictors of Bronchial Thermoplasty Response in Patients With Severe Refractory Asthma (BTR Study)
Acronym: BTR
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Cleveland Clinic (Other); National Jewish Health (Other); University of Arizona (Other); University of Chicago (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of Alabama at Birmingham (Other); Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0716- 201106118
Record Dates: First submitted 2010-06-21; First posted 2010-08-19 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA extraction, serum, plasma and sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe Asthma Patients: Severe asthma patients symptomatic despite high dose inhaled corticosteroid and long acting beta-agonist
  Interventions: Device: Alair system

INTERVENTIONS:
Device: Alair system — Bronchial thermoplasty

SUMMARY:
Clinical response, as defined by improvement in asthma quality of life, to bronchial thermoplasty in patients with severe refractory asthma can be predicted through the use of clinical, physiologic, biologic and imaging markers.

DETAILED DESCRIPTION:
Primary Aim To assess the relationship between baseline clinical, physiologic, biologic and imaging markers and response to bronchial thermoplasty, defined by improvement in asthma quality of life, in patients with severe refractory asthma.

Secondary Aims

1. To assess the relationship between baseline clinical, physiologic, biologic and imaging markers and response to bronchial thermoplasty, defined by reduction in severe exacerbations or healthcare utilization, in patients with severe refractory asthma.
2. To evaluate if baseline clinical, physiologic, biologic and imaging markers are related to safety of bronchial thermoplasty in patients with severe refractory asthma.
3. To evaluate and validate statistical models that predict response to bronchial thermoplasty in patients with severe refractory asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 or greater and less than 65
2. Subject has asthma and is taking regular maintenance medication for past 12 months that includes:

   * Inhaled corticosteroid (ICS) at a dosage greater than 1000μg beclomethasone per day or equivalent, AND long acting ß2-agonist (LABA) at a dosage of ≥100μg per day Salmeterol or equivalent.
   * Other asthma medications such as leukotriene modifiers, or anti-IgE, are acceptable (Subjects on Xolair® must have been on Xolair for greater than 1 year).
3. Asthma confirmed by: (a) b-agonist reversibility of FEV1 ≥ 12 % following 360mcg albuterol OR (b) methacholine FEV1 PC20 ≤ 8 mg/ml if not receiving an ICS or ≤ 16 mg/ml if receiving an ICS.
4. FEV1 ≥ 50% predicted pre-bronchodilator.
5. Asthma symptoms on at least two days or one night per week over the last 2 weeks.
6. Subject is a non-smoker for 1 year or greater (if former smoker, less than 10 pack years total smoking history).
7. Ability to undergo bronchoscopy in the opinion of the investigator.
8. Ability and willingness to provide informed consent.

Exclusion Criteria:

1. Asthma exacerbation (ED visit, hospitalization, course of increased systemic steroids, or urgent health care visit for asthma) during the prior four weeks.
2. Subject has 3 or more hospitalizations for exacerbations of asthma in the previous year or 1 or more ICU admission for asthma in the previous year.
3. Chronic oral steroid therapy greater than 30 mg per day
4. Subject has other respiratory diseases including interstitial lung disease, emphysema, cystic fibrosis, vocal cord dysfunction, mechanical upper airway obstruction, untreated obstructive sleep apnea, Churg-Strauss syndrome, cardiac dysfunction, and allergic bronchopulmonary aspergillosis (total IgE of >1000 Units/mL with positive specific IgE to aspergillus and evidence of central bronchiectasis) that in the opinion of the investigator would prevent participation in the trial or put the participant at risk by participation.
5. Subject has segmental atelectasis, lobar consolidation, significant or unstable pulmonary infiltrate, or pneumothorax, confirmed on x-ray.
6. Subject has clinically significant cardiovascular disease, including myocardial infarction, angina, cardiac dysrhythmia, conduction defect, cardiomyopathy, aortic aneurysm, or stroke.
7. Subject has uncontrolled hypertension (>200mm Hg systolic or >100mm Hg diastolic pressure).
8. Subject uses an internal or external pacemaker or cardiac defibrillator.
9. Chronic diseases (other than asthma) that in the opinion of the investigator would prevent participation in the trial or put the participant at risk by participation, e.g. chronic diseases of the lung (other than asthma), heart, liver, kidney, or nervous system, or immunodeficiency
10. History of cigarette smoking with > 10 pack years total
11. Use of investigative drugs or intervention trials in the 30 days prior to enrollment or during the duration of the study
12. Any condition or compliance issue which in the opinion of the investigator might interfere with participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject Population - Severe Refractory Asthma
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2010-08; Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Baseline predictors of response to bronchial thermoplasty defined by improvement in asthma quality of life, in patients with severe refractory asthma. | 12 months following last bronchial thermoplasty treatment
  To assess the relationship between baseline clinical, physiologic, biologic and imaging markers and response to bronchial thermoplasty, defined by improvement in asthma quality of life, in patients with severe refractory asthma.

SECONDARY OUTCOMES:
Baseline predictors of severe exacerbations | 12 months following last bronchial thermoplasty treatment
  To assess the relationship between baseline clinical, physiologic, biologic and imaging markers and response to bronchial thermoplasty, defined by reduction in severe exacerbations, in patients with severe refractory asthma.
Baseline predictors of healthcare utilization | 12 months following last bronchial thermoplasty treatment
  To assess the relationship between baseline clinical, physiologic, biologic and imaging markers and response to bronchial thermoplasty, defined by reduction in healthcare utilization, in patients with severe refractory asthma.
Baseline predictors of safety of bronchial thermoplasty | 12 months following last bronchial thermoplasty treatment
  To evaluate if baseline clinical, physiologic, biologic and imaging markers are related to safety of bronchial thermoplasty in patients with severe refractory asthma.
Predictive models of response to bronchial thermoplasty | 12 months following last bronchial thermoplasty treatment
  To evaluate and validate statistical models that predict response to bronchial thermoplasty in patients with severe refractory asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Castro, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - National Jewish Health, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Louisiana State University Health Sciences Center in New Orleans, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Samant M, Krings JG, Lew D, Goss CW, Koch T, McGregor MC, Boomer J, Hall CS, Schechtman KB, Sheshadri A, Peterson S, Erzurum S, DePew Z, Morrow LE, Hogarth DK, Tejedor R, Trevor J, Wechsler ME, Sam A, Shi X, Choi J, Castro M. Use of Quantitative CT Imaging to Identify Bronchial Thermoplasty Responders. Chest. 2024 Apr;165(4):775-784. doi: 10.1016/j.chest.2023.12.015. Epub 2023 Dec 18. PMID 38123124